CLINICAL TRIAL: NCT06842433
Title: The NUTRIOME Meal Study - a Data-driven Precision Nutrition Intervention Study Using Meal Responses
Brief Title: The NUTRIOME Study - a Data-driven Precision Nutrition Intervention
Acronym: NUTRIOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chalmers University of Technology (Other)
Collaborators: University of Oslo (Other); Wageningen University (Other); Polish Academy of Sciences (Other); Maastricht University (Other); German Cancer Research Center (Other); University of Copenhagen (Other); University of Oulu (Other); University College Dublin (Other)
Responsible Party: Principal Investigator, Rikard Landberg, Professor, Chalmers University of Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Nutriome
Record Dates: First submitted 2025-01-30; First posted 2025-02-24 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Control

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The dietary intervention of personalized dietary advice vs. general healthy diet will be blinded and matched for delivery of intervention and intensity.
  Wherever possible Care providers and researchers conducting the analysis (e.g., nurses drawing blood samples) will be blinded to the allocation of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- General healthy diet (Active Comparator): General healthy diet based on national health dietary guidelines.
  Interventions: Other: General healthy diet
- Personalized diet (Experimental): Personalized diet will be based on an algorithm considering the individuals' postprandial glucose, triglycerides and inflammation markers to each of the three study meals in the characterization phase (Phase I) matched with established knowledge about the effects of specific foods on such metabolic parameters
  Interventions: Other: Personalized diet

INTERVENTIONS:
Other: General healthy diet — General healthy diet based on national health dietary guidelines.
  Arms: General healthy diet
Other: Personalized diet — Personalized diet will be based on an algorithm considering the individuals' postprandial glucose, triglycerides and inflammation markers to each of the three study meals in the characterization phase (Phase I) matched with established knowledge about the effects of specific foods on such metabolic parameters.
  Arms: Personalized diet

SUMMARY:
The overall objective of this multi-center study is to use metabolic response data from different dietary challenges to develop personalized dietary advice. Effectiveness of this personalized dietary advice compared to a general healthy diet based on national dietary guidelines on markers of cardio-metabolic health will be tested.

A total of 120 men and women who meet all inclusion criteria and none of the exclusion criteria will be invited to participate. The study will be conducted at three sites: Chalmers University of Technology (Sweden), University of Wageningen (Netherlands), and University of Oslo (Norway), with 40 participants per site.The study is conducted in two parts. The first part, the characterization phase, is a three-way randomized, controlled cross-over design, featuring one-day meal tests with isocaloric meals containing different carbohydrate, fat and protein quantity as well as quality. Based on the metabolic response to the meal tests a personalized diet will be constructed. In the second part, the main intervention, effectiveness of this personalized dietary advice compared to a general healthy diet will be tested in a six week parallel group intervention study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 40 to 70 years
* Body mass index (BMI) 27-35 kg/m2
* Signed informed consent

Exclusion Criteria:

* History of diagnosed cardiovascular disease (e.g. stroke, heart disease)
* Diagnosed type 1 or type 2 diabetes
* Finger prick glucose test at screening indicating diabetes (fasting >6.9 mmol/L; non-fasting >11.0 mmol/L)
* Antibiotic use in the last 3 months
* Taking medication that can interfere with the planned outcome measures, as judged by the study physician (e.g. peroxisome proliferator-activated receptor-α [PPAR-α] or PPAR-γ agonists [fibrates], sulfonylureas, biguanides, α-glucosidase inhibitors, thiazolidinediones, repaglinide, nateglinide and insulin, chronic use of NSAIDs). Statins and hypertension medication are allowed if the medication regimen has been stable for the last three months
* Stomach and gastrointestinal conditions (e.g. Morbus Chron, Ulcerative colitis, irritable bowel syndrome, malabsorption, colostomy, bowel resection, gastric bypass surgery etc.)
* History of major gastrointestinal surgery
* Anaemia: Hb concentrations < 8.5 mmol/L for men and < 7.5 mmol/L for women
* Recent blood donation (within 2 months prior to the screening)
* Recent participation in another intervention study (within 2 months prior to the screening)
* Allergy or intolerance to medical skin adhesives
* Chronic or acute inflammatory conditions (e.g., rheumatoid arthritis, psoriatic arthritis)
* Autoimmune disorders
* Thyroid disorders
* Significant renal or liver dysfunction or chronic kidney or liver disease
* Known food allergies/intolerances to intervention foods or food products used in the study
* Following specific dietary regimen that could impact results or not suitable for the study design (e.g. vegetarian, vegan)
* Habitual tobacco consumption (e.g. smoking, use of snus, vaping)
* Alcohol intake ≥ 14 alcoholic beverages/week for women and ≥ 21 alcoholic beverages/week for men
* Current or planned pregnancy or lactating
* Other serious medical conditions that could interfere with participation or study outcomes
* Unable to sufficiently understand written and spoken national language (where the study centre is located) to provide written consent and understand information and instructions from the study personnel.
* Deemed unsuitable for participation in the trial, for any reason, as judged by the research physician or PI.
* Working at the division conducting the trial at any of the three study centres.
* Do not have a mobile phone that is suitable for the use of a research app.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Glucose postprandial | 6 weeks
  Difference between groups in postprandial glucose in response to a mixed meal tolerance test.
Triglycerides postprandial | 6 weeks
  Difference between groups in postprandial triglycerides in response to a mixed meal tolerance test.
Interleukin-6 postprandial | 6 weeks
  Difference between groups in postprandial interleukin-6 in response to a mixed meal tolerance test.

SECONDARY OUTCOMES:
Inflammatory markers in blood | 6-hour meal test
  Differences in immunological responses (such as cytokines, lipopolysaccharides, GlycA) between test meals in the characterization phase of the study.
Appetite | 6-hour meal test
  Differences in self-reported appetite measured using a visual analogue scale between test meals in the characterization phase of the study.
Gut microbiome | 6-hour meal test
  Differences in fecal microbiome between test meals in the characterization phase of the study.
Metabolome | 6-hour meal test
  Differences in metabolome (plasma, urine and feces) between test meals in the characterization phase of the study.
Lipid metabolism | 6-hour meal test
  Differences in lipid metabolism between test meals in the characterization phase of the study.
Glycemic variability | 4 weeks
  Differences in glycemic variability across the different meals and the OGTT throughout the characterization phase of the study.
Gastrointestinal hormones | 6-hour meal test
  Release of gastrointestinal hormones (such as GLP-1, CCK) in response to the test meals in the characterization phase of the study.
Fecal proteome | 6-hour meal test
  Differences in fecal proteome between test meals in the characterization phase of the study.
PBMC Transcriptome | 6-hour meal test
  Differences in peripheral blood mononuclear cell gene expression between test meals in the characterization phase of the study.
PBMC Epigenome | 6-hour meal test
  Differences in peripheral blood mononuclear cell epigenome between test meals in the characterization phase of the study.
PBMC Immunometabolism | 6-hour meal test
  Differences in peripheral blood mononuclear cell immunometabolism between test meals in the characterization phase of the study.
Metabolome | 6 weeks
  Difference in metabolome (plasma, urine and feces) between personalized diet and general healthy diet in the intervention phase of the study.
PBMC Epigenome | 6 weeks
  Difference in peripheral blood mononuclear cell epigenome between personalized diet and general healthy diet in the intervention phase of the study.
PBMC Transcriptome | 6 weeks
  Difference in peripheral blood mononuclear cell transcriptome between personalized diet and general healthy diet in the intervention phase of the study.
PBMC Immunometabolism | 6 weeks
  Difference in peripheral blood mononuclear cell immunometabolism between personalized diet and general healthy diet in the intervention phase of the study.
Fecal proteome | 6 weeks
  Difference in fecal proteome between personalized diet and general healthy diet in the intervention phase of the study.
Gut microbiome | 6 weeks
  Difference in fecal microbiome between personalized diet and general healthy diet in the intervention phase of the study.
Inflammatory markers in blood | 6 weeks
  Differences in immunological responses (such as cytokines, lipopolysaccharides, GlycA) to mixed meal tolerance tests between personalized diet and general healthy diet in the intervention phase of the study.
Glycemic variability | 6 weeks
  Differences in glycemic variability between personalized diet and general healthy diet in the intervention phase of the study.
Data-driven prediction of response to intervention | 6 weeks
  Data-driven prediction of primary and other outcomes to personalized diet vs. general healthy diet using metabolome, gut microbiome, epigenome, transcriptome, proteome, immunometabolism, health measures, lifestyle and metabolic markers as determinants.

OTHER OUTCOMES:
Dietary biomarkers | 6-hour meal test and 6 week intervention
  Exploratory analysis of blood, urine and feces to find potential biomarkers reflecting dietary intake in the characterization and intervention phase of the study.
Responsivness to diet | 6-hour test meal and 6 week intervention
  Exploration of underlying mechanisms behind response/non-response to personalized and general healthy diet using data from both the characterization phase (meal test) and the primary 6-week intervention.
Gastric emptying | 6-hour test meal
  Gastric emptying will be assessed by breath test at one of the test meals in a sub-group of participants (Swedish and Norwegian site).
Gastric passage time | 6-hour meal test and 6 week intervention
  Gastric passage time will be assessed using the blue dye method.

CONTACTS AND LOCATIONS:
Locations (3):
- Wageningen University and Research, Human research unit, Wageningen, Netherlands
- Department of nutrition, University of Oslo, Oslo, Norway
- University of Gothenburg, Department of Internal medicin and Clinical nutrition, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided